CLINICAL TRIAL: NCT00334438
Title: A Phase I Study Evaluating Combined Zevalin (Ibritumomab Tiuxetan) and Valcade (Bortezomib) in Relapsed/Refractory Low-Grade or Follicular B-Cell and Mantle Cell Lymphoma
Brief Title: Bortezomib, Rituximab, and Yttrium Y 90 Ibritumomab Tiuxetan in Treating Patients With Relapsed or Refractory Low-Grade, Follicular, or Mantle Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0525; CDR0000550130 (Other: PDQ number)
Record Dates: First submitted 2006-06-06; First posted 2006-06-07 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent small lymphocytic lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Bortezomib; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zevalin + Velcade Single Arm Study (Other): Zevalin (Ibritumomab Tiuxetan) and Velcade (Bortezomib)
  Interventions: Biological: rituximab; Drug: bortezomib; Radiation: yttrium Y 90 ibritumomab tiuxetan; Radiation: Indium 111 ibritumomab tiuxetan

INTERVENTIONS:
Biological: rituximab — 250mg/m2, IV, Days 1 and 8
  Other Names: Rituxan
Drug: bortezomib — dose escalation 1.0, 1.3, or 1.5, IVP; Days 4, 8, 11, 15
  Other Names: Velcade
Radiation: yttrium Y 90 ibritumomab tiuxetan — Dose dependant upon platelet count (0.4mCi/kg) not to exceed 32mCi; Day 8
Radiation: Indium 111 ibritumomab tiuxetan — 5cmCi; IV day 1

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, and radiolabeled monoclonal antibodies, such as yttrium Y 90 ibritumomab tiuxetan, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them without harming normal cells. Giving bortezomib together with rituximab and yttrium Y 90 ibritumomab tiuxetan may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of bortezomib when given together with rituximab and yttrium Y 90 ibritumomab tiuxetan in treating patients with relapsed or refractory low-grade, follicular, or mantle cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of bortezomib in combination with rituximab and yttrium Y 90 ibritumomab tiuxetan in patients with relapsed or refractory low-grade, follicular B-cell, or mantle cell non-Hodgkin's lymphoma.
* Determine the dose-limiting toxicity of this regimen in these patients.

Secondary

* Determine the response rate in patients treated with this regimen.

OUTLINE: This is a multicenter, open-label, nonrandomized, dose-escalation study of bortezomib.

Patients receive rituximab IV over 4 hours followed by indium In 111 ibritumomab tiuxetan IV over 10 minutes on day 1 to assess biodistribution. Patients without altered biodistribution receive rituximab IV over 4 hours followed by yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day 8. Patients also receive bortezomib IV over 3-5 seconds on days 4, 8, 11, and 15.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Additional patients may be treated at the MTD.

After completion of study treatment, patients are followed every 3 months for 18 months and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed low-grade, follicular B-cell, or mantle cell non-Hodgkin's lymphoma

  * Bone marrow biopsy required for pretreatment evaluation

    * Unilateral bone marrow biopsy allowed
    * Core biopsies allowed if they contain adequate tissue for primary diagnosis and immunophenotyping
* Relapsed or refractory disease as defined by disease progression after initial complete response (CR) or failure to achieve CR
* No bone marrow involvement ≥ 25% within the past 30 days
* No pleural effusion or significant ascites
* No active CNS involvement

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* AST ≤ 2.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 2.5 times ULN
* Creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Hepatitis B surface antigen negative
* No current infection with hepatitis B virus
* No HIV positivity
* No neuropathy or neuropathic pain ≥ grade 2
* No history of allergic reaction to boron or mannitol
* No active serious infection or medical or psychiatric illness that would preclude study therapy
* No other malignancy within the past 5 years except for the following:

  * Basal cell or squamous cell carcinoma of the skin that has been completely resected
  * In situ malignancy that has been completely resected
  * T1-T2a, N0, M0 prostate cancer treated with a prostatectomy or radiotherapy within the past 2 years with an undetectable PSA level
* No other condition, including any of the following:

  * Myocardial infarction within the past 6 months
  * New York Heart Association class III-IV heart failure
  * Uncontrolled angina
  * Severe uncontrolled ventricular arrhythmias
  * Electrocardiographic evidence of acute ischemia or active conduction system abnormalities

PRIOR CONCURRENT THERAPY:

* Recovered from all prior therapy
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C), radiotherapy, or surgical resection of malignancy

  * No limitations on the number of prior therapies
* More than 4 weeks since prior major surgery
* More than 14 days since prior filgrastim (G-CSF) or sargramostim (GM-CSF)
* More than 14 days since prior and no other concurrent investigational agents

  * Concurrent participation in a nontreatment study allowed
* No prior radioimmunotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-07; Primary Completion 2008-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of bortezomib | 2 years
Dose-limiting toxicity | 8 weeks

SECONDARY OUTCOMES:
Response rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Shea, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina